CLINICAL TRIAL: NCT03642574
Title: Cumulative Live Birth Rate With eSET After Preimplantation DNA Methylation Test (PIMT) in ART
Brief Title: Preimplantation DNA Methylation Test (PIMT) in ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Zi-Jiang (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor-Investigator, Chen Zi-Jiang, Professor, Shandong University
Organization: Shandong University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIMT
Record Dates: First submitted 2018-08-16; First posted 2018-08-22 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: DNA Methylation
Keywords: Preimplantation Methylome Screening; Preimplantation Genetic Screening; single embryo transfer; cumulative live birth rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PIMT methylation (Experimental): Subjects will have blastocyst biopsy and whole genome DNA methylation sequencing done with 2 or 7 good-quality embryos on Day 5 to 7. Principle of freeze-all and single thawed blastocyst transfer will be applied. Only embryos with euploid chromosome will be transfered to the uterus. The outcome of all euploids transfers within 1 year will be followed up. During study, every subject will have at most one live birth.
  Interventions: Procedure: CNV

INTERVENTIONS:
Procedure: CNV — Embryo with euploid chromosome will transfer to uterus. The order of transfer is accroding to morphological grade.

SUMMARY:
The purpose of this clinical trial is to determine the safety and effect of methylation level of DNA methylation in embryos on the outcome of assisted reproductive technology (ART) during blastocyst embryo screening. Subjects with blastocysts on day 5-7 of embryo culture will be biopsied. A Freeze-all strategy and a single frozen blastocyst transfer will be performed till all study-specific embryos have been transferred. Then whole genome bisulfate sequencing will be performed on all cells that obtained from biopsy.

DETAILED DESCRIPTION:
The purpose of this clinical trial is to determine the safety and affect of DNA methylation level on ART. Subjects with blastocysts on day 5-7 of embryo culture will be biopsied. A Freeze-all strategy and a single frozen blastocyst transfer will be performed till all study-specific embryos have been transferred. Then whole genome bisulfate sequencing will be performed on all cells that obtained from biopsy. The investigators will perform whole genome DNA methylation sequence for two to seven blastocysts from one couple. The methylation level and genomic copy number variation will be analyzed by using the methylome data. Embryos with aneuploid chromosomes will be rejected for embryo transfer to uterus. The study will examine which kind of methylation level can produce the best clinical outcome for ART. Biopsied cells will perform with preimplnatation DNA methylation test (PIMT). DNA methylation level and chromosome copy number variation will be calculated by using whole genome DNA methylation sequencing data. As we do not kown which kind of methylation state can produce the best outcome in ART practice. This study will try to find a standard of selection embryos according to DNA methylation information. Under current stage, the selection of embryo is according to chromosome copy number. The embryo selection will not consider DNA methylation information for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are participating in preimplantation screening with PGS indications,defined as maternal age above 38 years, repeated implantation failure (RIF) usually defined as three or more transfers of morphologically high-quality embryos without the establishment of pregnancy, recurrent miscarriage (RM) in patients with normal karyotypes (usually at least three previous consecutive miscarriages) and severe male factor infertility (usually defined as abnormal semen parameters).
2. Women who obtain 2 or more good-quality blastocysts that defined as morphological score of inner cell mass B or A, trophectoderm C or better, and grade 4 or better on Day five of embryo culture will be randomized.

Exclusion Criteria:

1. Women with a uterine cavity abnormality, such as a uterine congenital malformation (uterus unicornate, bicornate, or duplex); untreated uterine septum, adenomyosis, submucous myoma, or endometrial polyp(s); or with history of intrauterine adhesions.
2. Women with untreated hydrosalpinx.
3. Women who use donated oocytes or sperm to achieve pregnancy.
4. Women with contraindication for assisted reproductive technology or for pregnancy, such as poorly controlled Type I or Type II diabetes; undiagnosed liver disease or dysfunction (based on serum liver enzyme testing); renal disease or abnormal serum renal function; significant anemia; history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident; uncontrolled hypertension, known symptomatic heart disease; history of or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma; undiagnosed vaginal bleeding.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The effect of DNA methylation level on live birth rate | 22 months
  The rate of live birth at different methylation level will be calculated. Live birth is defined as the delivery of any viable infant at 28 weeks or more of gestation, and cumulative live birth rate is calculated by dividing the number of women achieving live birth after transfers (up to 3 transfers of single blastocycst within 1 year).

SECONDARY OUTCOMES:
The effect of DNA methylation level on pregnant rate, pregnant loss rate. | 22 months
  The rate of pregnant and pregnant loss at different methylation level will be calculated. Pregnancy loss refers to a complete spontaneous abortion or a nonviable pregnancy before 28 weeks of gestation.
Duration of pregnancy | 22 months
  The time from the first day of last menstrual period to the day of delivery.
Birth weight | 22 months
  Weight of newborns at delivery.
Cumulative incidence of maternal complications during whole | 22 months
  Number of pregnancies with complications / number of pregnancies over (up to) 3 transfers within 1 year;
Cumulative incidence of neonatal complications during whole | 22 months
  Number of live births with neonatal complications / number of live births over (up to)3 transfers within 1 year
Number of embryo transfers to achieve live birth | 22 months
  Number of embryo transfers the patients have gone through to achieve live birth.

OTHER OUTCOMES:
Clinical pregnancy rate after the first transfer | 4 months
  Number of women with clinical pregnancies after the first transfer / number of women.
Pregnancy loss rate after the first transfer | 9 months
  Number of pregnancy losses / number of clinical pregnancies after the first transfer .
Live birth rate after the first transfer | 12 months
  Number of women with live births after the first transfer / number of women.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brezina PR, Kutteh WH. Clinical applications of preimplantation genetic testing. BMJ. 2015 Feb 19;350:g7611. doi: 10.1136/bmj.g7611. PMID 25697663
- [Background] Hassold T, Chen N, Funkhouser J, Jooss T, Manuel B, Matsuura J, Matsuyama A, Wilson C, Yamane JA, Jacobs PA. A cytogenetic study of 1000 spontaneous abortions. Ann Hum Genet. 1980 Oct;44(2):151-78. doi: 10.1111/j.1469-1809.1980.tb00955.x. PMID 7316468
- [Background] Dahdouh EM, Balayla J, Audibert F; Genetics Committee; Wilson RD, Audibert F, Brock JA, Campagnolo C, Carroll J, Chong K, Gagnon A, Johnson JA, MacDonald W, Okun N, Pastuck M, Vallee-Pouliot K. RETIRED: Technical Update: Preimplantation Genetic Diagnosis and Screening. J Obstet Gynaecol Can. 2015 May;37(5):451-63. doi: 10.1016/s1701-2163(15)30261-9. PMID 26168107
- [Background] Kalousek DK, Pantzar T, Tsai M, Paradice B. Early spontaneous abortion: morphologic and karyotypic findings in 3,912 cases. Birth Defects Orig Artic Ser. 1993;29(1):53-61. No abstract available. PMID 8280893
- [Background] Smith ZD, Meissner A. DNA methylation: roles in mammalian development. Nat Rev Genet. 2013 Mar;14(3):204-20. doi: 10.1038/nrg3354. Epub 2013 Feb 12. PMID 23400093
- [Background] Jones PA. Functions of DNA methylation: islands, start sites, gene bodies and beyond. Nat Rev Genet. 2012 May 29;13(7):484-92. doi: 10.1038/nrg3230. PMID 22641018
- [Background] Jiang L, Zhang J, Wang JJ, Wang L, Zhang L, Li G, Yang X, Ma X, Sun X, Cai J, Zhang J, Huang X, Yu M, Wang X, Liu F, Wu CI, He C, Zhang B, Ci W, Liu J. Sperm, but not oocyte, DNA methylome is inherited by zebrafish early embryos. Cell. 2013 May 9;153(4):773-84. doi: 10.1016/j.cell.2013.04.041. PMID 23663777
- [Background] Li G, Yu Y, Fan Y, Li C, Xu X, Duan J, Li R, Kang X, Ma X, Chen X, Ke Y, Yan J, Lian Y, Liu P, Zhao Y, Zhao H, Chen Y, Sun X, Liu J, Qiao J, Liu J. Genome wide abnormal DNA methylome of human blastocyst in assisted reproductive technology. J Genet Genomics. 2017 Oct 20;44(10):475-481. doi: 10.1016/j.jgg.2017.09.001. Epub 2017 Sep 6. PMID 29037989
- [Background] Schieve LA, Meikle SF, Peterson HB, Jeng G, Burnett NM, Wilcox LS. Does assisted hatching pose a risk for monozygotic twinning in pregnancies conceived through in vitro fertilization? Fertil Steril. 2000 Aug;74(2):288-94. doi: 10.1016/s0015-0282(00)00602-6. PMID 10927046
- [Background] Fiorentino F, Biricik A, Bono S, Spizzichino L, Cotroneo E, Cottone G, Kokocinski F, Michel CE. Development and validation of a next-generation sequencing-based protocol for 24-chromosome aneuploidy screening of embryos. Fertil Steril. 2014 May;101(5):1375-82. doi: 10.1016/j.fertnstert.2014.01.051. Epub 2014 Mar 6. PMID 24613537
- [Background] Shi Y, Sun Y, Hao C, Zhang H, Wei D, Zhang Y, Zhu Y, Deng X, Qi X, Li H, Ma X, Ren H, Wang Y, Zhang D, Wang B, Liu F, Wu Q, Wang Z, Bai H, Li Y, Zhou Y, Sun M, Liu H, Li J, Zhang L, Chen X, Zhang S, Sun X, Legro RS, Chen ZJ. Transfer of Fresh versus Frozen Embryos in Ovulatory Women. N Engl J Med. 2018 Jan 11;378(2):126-136. doi: 10.1056/NEJMoa1705334. PMID 29320646
- [Background] Chen ZJ, Shi Y, Sun Y, Zhang B, Liang X, Cao Y, Yang J, Liu J, Wei D, Weng N, Tian L, Hao C, Yang D, Zhou F, Shi J, Xu Y, Li J, Yan J, Qin Y, Zhao H, Zhang H, Legro RS. Fresh versus Frozen Embryos for Infertility in the Polycystic Ovary Syndrome. N Engl J Med. 2016 Aug 11;375(6):523-33. doi: 10.1056/NEJMoa1513873. PMID 27509101